CLINICAL TRIAL: NCT05441527
Title: Use of Two Dissolvable Therapeutics Under Removable Partial Dentures: Reported Effects on Denture Comfort, Retention, and Dry Mouth Conditions
Brief Title: Use of Two Dissolvable Therapeutics Under Removable Partial Dentures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iowa (Other)
Responsible Party: Principal Investigator, Robert Bowers, Assistant Professor, University of Iowa
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 202104384
Record Dates: First submitted 2022-06-28; First posted 2022-07-01 (Actual); Results first posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Edentulous Jaw; Edentulous Mouth
MeSH Terms: conditions — Jaw, Edentulous; Mouth, Edentulous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- MI Paste, then, Biotene Dry Mouth Gel (Experimental): Subjects in this arm will use 1 milliliter of MI Paste daily for 7 days. Then, the subjects in this arm will use 1 milliliter of Biotene Dry Mouth gel daily for 7 days. There will be no wash-out period between the two products.
  Interventions: Device: MI Paste, then, Biotene Dry Mouth Gel
- Biotene Dry Mouth Gel, then, MI Paste (Experimental): Subjects in this arm will use 1 milliliter of Biotene Dry Mouth gel for 7 days. Then, the subjects in this arm will use 1 milliliter of MI Paste for 7 days. There will be no wash-out period between the two products.
  Interventions: Device: Biotene Dry Mouth Gel, then, MI Paste

INTERVENTIONS:
Device: MI Paste, then, Biotene Dry Mouth Gel — 1 milliliter of product will be applied daily to the intaglio (i.e., underside) of the patient's removable prosthesis and seated intraorally.
  Arms: MI Paste, then, Biotene Dry Mouth Gel
Device: Biotene Dry Mouth Gel, then, MI Paste — 1 milliliter of product will be applied daily to the intaglio (i.e., underside) of the patient's removable prosthesis and seated intraorally.
  Arms: Biotene Dry Mouth Gel, then, MI Paste

SUMMARY:
Older removable denture wearing adults suffer from a complex set of oral health challenges, with relatively few solutions identified at this time. This is substantiated by statistics concerning the geriatric population on the correlation of poor oral health and the degradation of an individual's overall quality of life. The most recent National Health and Nutrition Examination Survey data found that 1 in 8 U.S. adults over the age of 65 are completely edentulous. A shift from complete edentulism to partial edentulism was also seen in this survey data, as the average individual over 65 had only 21 teeth remaining. Thus, partial edentulism remains a significant burden on seniors as well.

Clearly, there exists both a great need and desire for improved implementation of proven oral-health strategies among this population, as well as the development of new preventive interventions and minimally invasive treatment strategies beyond traditional denture adhesive products.

This proposed clinical trial intends to investigate two such potential treatment aids. In follow-up from our recent pilot study investigating MI Paste's application on the intaglio of complete dentures, in which our current findings have shown that the use of MI Paste can predictably increase the buffering capacity of a patient's saliva, our current proposal targets to further increase the study's sample size to improve the statistical power regarding subjective patient reports.

The primary aims of this proposed study are to collect further data on how MI Paste affects patients' subjective evaluations of the comfort and retention of their denture, as well as dry mouth symptoms in patients reporting xerostomia.

Furthermore, this study will include a second therapeutic intervention, Biotene Dry Mouth Gel (OTC), which will provide an additional contrast variable involving patient preferences regarding therapeutics under their removable prostheses. We hypothesize that the use of both therapeutics underneath removable dentures will provide added retention and stability to the prosthesis on patient reports, further coinciding with improved evaluations of comfort and function. Additionally, we hypothesize that the subjective improvements in patients self-reporting xerostomia will be of a statistically greater magnitude than those noticed by patients with normal salivary function, as xerostomia has been associated with increased denture discomfort in past literature.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-99
* Patients with a removable prosthesis (e.g., partial denture, complete denture)
* Removable prosthesis must have been made at the University of Iowa College of Dentistry's Department of Family Dentistry clinic within the past 10 years.

Exclusion Criteria:

* Casein (i.e., protein found in milk or other dairy products) allergy
* Lactose intolerance
* Multiple food or cosmetic ingredient allergies in their health history
* Ill-fitting dentures that need to be remade or relined

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2022-06-30 (Actual); Primary Completion 2024-05-27 (Actual); Study Completion 2024-05-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Bowers, DDS, Principal Investigator — University of Iowa College of Dentistry
Locations (1):
- University of Iowa College of Dentistry, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Biotene, Then MI Paste: Subjects in this arm will use 1 milliliter of Biotene Dry Mouth gel for 7 days. After no wash-out period, the subject will switch to 1 milliliter of MI Paste for 7 days.
  1 milliliter of product will be applied daily to the intaglio (i.e., underside) of the patient's removable prosthesis and seated intraorally.
- MI Paste, Then Biotene: Subjects in this arm will use 1 milliliter of MI Paste for 7 days. After no wash-out period, the subject will switch to 1 milliliter of Biotene for 7 days.
  1 milliliter of product will be applied daily to the intaglio (i.e., underside) of the patient's removable prosthesis and seated intraorally.
Period: First Intervention (7 Days)
Arm/Group | Biotene, Then MI Paste | MI Paste, Then Biotene
Started | 29 | 24
Received Intervention | 29 | 24
Completed | 29 | 24
Not Completed | 0 | 0
Period: Second Intervention (7 Days)
Arm/Group | Biotene, Then MI Paste | MI Paste, Then Biotene
Started | 29 | 24
Completed | 29 | 23
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Biotene, Then MI Paste | MI Paste, Then Biotene | Total
Number analyzed (Participants) | 29 | 24 | 53
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 11 | 19
  >=65 years | 21 | 13 | 34
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 13 | 31
  Male | 11 | 11 | 22
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 29 | 24 | 53

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Patient Comfort for as Assessed by Numerical Scale.
Description: Comfort will be measured on a numerical scale of 0 to 10, where 0 is very dissatisfied and 10 is very satisfied.
Time Frame: Baseline, 1 week
Population: The average of patient comfort was calculated before the intervention. Then, after the intervention, the average of patient comfort was assessed again, and the difference between pre- and post-treatment is reported in alignment with the outcome of change from baseline in patient comfort for as assessed by numerical scale.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Biotene: Subjects in this arm will use either 1 milliliter of Biotene Dry Mouth gel for either the first 7 days of the study or the last 7 days of the study.
- MI Paste: Subjects in this arm will use either 1 milliliter of MI Paste for the first 7 days of the study or for the last 7 days of the study.
Arm/Group | Biotene | MI Paste
Number analyzed (Participants) | 52 | 53
units on a scale | 0.99 (1.64) | 1.16 (1.70)

2. Primary Outcome: Change From Baseline in Retention as Assessed by Numerical Scale.
Description: Retention will be measured on a numerical scale of 0 to 10, where 0 is very dissatisfied and 10 is very satisfied.
Time Frame: Baseline, 1 week
Population: The average of retention was calculated before the intervention. Then, after the intervention, the average of retention was assessed again, and the difference between pre- and post-treatment is reported in alignment with the outcome of change from baseline retention for as assessed by numerical scale.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Biotene Dry Mouth Gel: Subjects in this arm will use 1 milliliter of Biotene Dry Mouth Gel for either the first 7 days of the study or the last 7 days of the study.
- MI Paste: Subjects in this arm will use 1 milliliter of MI Paste for either the first 7 days of the study or the last 7 days of the study.
Arm/Group | Biotene Dry Mouth Gel | MI Paste
Number analyzed (Participants) | 52 | 53
units on a scale | 0.56 (1.85) | 0.97 (1.39)

ADVERSE EVENTS:
Time Frame: 2 weeks
Groups:
- MI Paste: Subjects in this arm will use 1 milliliter of MI Paste gel for either the first 7 days of the study or the last 7 days of the study.
Arm/Group | Biotene Dry Mouth Gel | MI Paste
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/53
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/53
Other Adverse Events (participants affected / at risk) | 0/52 | 0/53

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-05-28): https://cdn.clinicaltrials.gov/large-docs/27/NCT05441527/Prot_SAP_000.pdf